CLINICAL TRIAL: NCT05698342
Title: Tissue-resident Memory T Cells Expression in Melasma
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Clinical and research professor in Dermatology, Universidad Autonoma de San Luis Potosí
Other Study IDs: 81-21
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Melasma
Keywords: blimp-1; runx-3; transcription factors; tissue-resident memory T cells
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — two- 3 mm punch skin biopsies from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Melasma mMASI 7: Female patients with melasma mMASI at least 7

SUMMARY:
The treatment of melasma and the maintenance of depigmentation represent a challenge due to its frequent recurrences. Pathophysiological mechanisms and factors have been linked to melasma such as inflammation, sun exposure, increased CD4+ T lymphocytic infiltrate and IL-17 in damaged skin. Tissue-resident memory T cells (Trm), derived from naïve T lymphocytes, are associated with the recurrence of lesions at the same sites but they have not been described in melasma. This a Cross-sectional, prospective analytical study. 20 female patients, 18 to 55 years of age, with diagnosis of melasma and mMASI score of at least 7, at least 1-year duration, lesional and perilesional skin biopsies were taken for PCR and DIF. The objective is to determine the transcription factors of Trm cells in malar melasma.

DETAILED DESCRIPTION:
Melasma is a common, acquired pigmentary disorder characterized by chronic and relapsing hypermelanosis on sun-exposed areas that causes significant emotional and psychosocial impact in patients mainly in women with Fitzpatrick III-V phototypes. The treatment of melasma and the maintenance of depigmentation represents a challenge due to its frequent recurrences.

Different pathophysiological mechanisms and factors have been linked to melasma such as inflammation, sun exposure, increased CD4+ T lymphocytic infiltrate and IL-17 in damaged skin. In pathologies such as vitiligo and psoriasis, tissue-resident memory T cells (Trm), derived from naïve T lymphocytes, are associated with the recurrence of lesions at the same sites. These cells have a specific profile of transcription factors (Runx3+, Notch+, Blimp1+) and CD69 + CD103 + markers. These cells have not been described in melasma.

Objective: to determine the transcription factors of Trm cells in malar melasma. This is a Cross-sectional, prospective analytical study. 20 female patients, 18 to 55 years of age, with diagnosis of melasma and mMASI score of at least 7, at least1 year duration, and no treatment in the last 4 weeks, were included. Lesional and perilesional skin biopsies were taken for PCR and DIF. The presence of trm cells has not been described or studied in melasma where there is recurrence of the dermatosis in the same site, it is essential to understand its pathogenesis in order to address directed future therapies targeting these cells that may related to the disease.

ELIGIBILITY:
Inclusion Criteria:

female patients with malar melasma, healthy volunteers 18 years of age and older, without previous treatment or photoprotection measures within the previous 4 weeks, who had at least 7 Modified Melasma Activity and Severity Index (mMASI) score

Exclusion Criteria:

* Exclusion criteria were pregnancy or nursing, menopause, coexistence of other pigmentation conditions, heat exposure, regular exer- cise, diet restriction, consumption of food supplements or any type of drugs (including anti-inflammatories and hormonal treatments) within the previous 2 months, and women who had given birth within 1 year

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: female patients with malar melasma, healthy volunteers 18 years of age and older, without previous treatment or photoprotection measures within the previous 4 weeks, who had at least 7 Modified Melasma Activity and Severity Index (mMASI) score
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Tissue-resident memory T cells | up to 1 year
  To determine the difference in the levels of transcription factors of TRM cells in lesional skin and perilesional skin of patients with melasma

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Filoni A, Mariano M, Cameli N. Melasma: How hormones can modulate skin pigmentation. J Cosmet Dermatol. 2019 Apr;18(2):458-463. doi: 10.1111/jocd.12877. Epub 2019 Feb 18. PMID 30779300
- [Result] Hernandez-Barrera R, Torres-Alvarez B, Castanedo-Cazares JP, Oros-Ovalle C, Moncada B. Solar elastosis and presence of mast cells as key features in the pathogenesis of melasma. Clin Exp Dermatol. 2008 May;33(3):305-8. doi: 10.1111/j.1365-2230.2008.02724.x. PMID 18419607
- [Result] Rodriguez-Arambula A, Torres-Alvarez B, Cortes-Garcia D, Fuentes-Ahumada C, Castanedo-Cazares JP. CD4, IL-17, and COX-2 Are Associated With Subclinical Inflammation in Malar Melasma. Am J Dermatopathol. 2015 Oct;37(10):761-6. doi: 10.1097/DAD.0000000000000378. PMID 26381025
- [Result] Lee HC, Thng TG, Goh CL. Oral tranexamic acid (TA) in the treatment of melasma: A retrospective analysis. J Am Acad Dermatol. 2016 Aug;75(2):385-92. doi: 10.1016/j.jaad.2016.03.001. Epub 2016 May 17. PMID 27206758
- [Result] Tokura Y, Phadungsaksawasdi P, Kurihara K, Fujiyama T, Honda T. Pathophysiology of Skin Resident Memory T Cells. Front Immunol. 2021 Feb 3;11:618897. doi: 10.3389/fimmu.2020.618897. eCollection 2020. PMID 33633737
- [Result] Watanabe R, Gehad A, Yang C, Scott LL, Teague JE, Schlapbach C, Elco CP, Huang V, Matos TR, Kupper TS, Clark RA. Human skin is protected by four functionally and phenotypically discrete populations of resident and recirculating memory T cells. Sci Transl Med. 2015 Mar 18;7(279):279ra39. doi: 10.1126/scitranslmed.3010302. PMID 25787765
- [Result] Zou Y, Yuan H, Zhou S, Zhou Y, Zheng J, Zhu H, Pan M. The Pathogenic Role of CD4+ Tissue-Resident Memory T Cells Bearing T Follicular Helper-Like Phenotype in Pemphigus Lesions. J Invest Dermatol. 2021 Sep;141(9):2141-2150. doi: 10.1016/j.jid.2021.01.030. Epub 2021 Mar 16. PMID 33741391
- [Result] Fraczek A, Owczarczyk-Saczonek A, Placek W. The Role of TRM Cells in the Pathogenesis of Vitiligo-A Review of the Current State-Of-The-Art. Int J Mol Sci. 2020 May 18;21(10):3552. doi: 10.3390/ijms21103552. PMID 32443482
- [Result] Adachi T, Kobayashi T, Sugihara E, Yamada T, Ikuta K, Pittaluga S, Saya H, Amagai M, Nagao K. Hair follicle-derived IL-7 and IL-15 mediate skin-resident memory T cell homeostasis and lymphoma. Nat Med. 2015 Nov;21(11):1272-9. doi: 10.1038/nm.3962. Epub 2015 Oct 19. PMID 26479922